CLINICAL TRIAL: NCT04342039
Title: Epigenetic Health Benefits of Budesonide
Acronym: Project Ace
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Genome British Columbia (Industry); Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Principal Investigator, Christopher Carlsten, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H20-00414
Record Dates: First submitted 2020-03-09; First posted 2020-04-10 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Epigenetic Effects of Intranasal Steroids; Environmental Exposure
Keywords: Controlled Human Exposure Study; Budesonide Nasal Spray; Epigenetics; Gene Expression; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: Participants will visit our lab for 2 trial cycles (each cycle involves one arm):
  1) Budesonide, and 2) placebo. Within each cycle, there are periods with and without pollution exposure, so there is a secondary comparison of pre- versus post-pollution exposure.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Visually indistinguishable placebo and budesonide nasal sprays will be coded by research staff not connected to the study and pre-packaged for participants. All assays will be performed by personnel who do not know the exposure conditions of individual samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will use a placebo nasal spray before being exposed to a series of allergen and pollution challenges.
  Interventions: Other: Placebo
- Budesonide nasal (Active Comparator): Participants will use budesonide nasal spray before being exposed to a series of allergen and pollution challenges.
  Interventions: Drug: Budesonide Nasal

INTERVENTIONS:
Drug: Budesonide Nasal — budesonide 64 mcg/spray; 2 sprays each nostril once daily on days as indicated in the timeline
  Other Names: Rhinocort
  Arms: Budesonide nasal
Other: Placebo — 2 sprays each nostril daily on days as indicated in the timeline
  Arms: Placebo

SUMMARY:
Around 40% of the world's population is now impacted by allergic disease and this figure continues to rise. It is now understood that allergic disease arises from complex interactions between genetic and environmental factors. Exposure to allergens such as dust mites and pollen, as well as air pollutants such as diesel exhaust particulates, can alter the ability of critical genes to be expressed appropriately, a process known as epigenetic modification. The epigenetic modifications induced by allergens and pollutants appears to be reversible, thus providing a mechanism by which allergic disease can be treated. Budesonide (Rhinocort®) is a corticosteroid nasal spray commonly used to treat allergy symptoms. While the anti- inflammatory and other pharmacological aspects of budesonide are well understood, recent studies have suggested that budesonide may also work by reversing the epigenetic modifications caused by allergen exposure, although this has not been examined in the context of real-world exposures in humans.

This study aims to harness the power of epigenetic analysis to determine whether the epigenetic landscape in patients suffering from allergic disease can be modified by the administration of budesonide. It will fill critical gaps in understanding of epigenetic effects and provide information to examine the connection between environmental impacts and treatment effects. The research will expand the mechanistic understanding of the therapeutic effects of budesonide for relief of nasal rhinitis symptoms and may reveal new mechanisms that could improve treatment of allergies or pollution exposure, or serve as a tool for evaluating future therapies. If this venture is successful, it will serve as a model for studying and optimizing the epigenetic effects of other treatments and other diseases.

DETAILED DESCRIPTION:
To test this, the investigators have planned for two treatment trials where participants will act as both the control and tester (crossover design method). Participants will be provided a randomized treatment order of either 1) Budesonide (Rhinocort) or 2) placebo (no medication) nasal spray for the treatment trial. Participants will go through a series of nasal sampling, symptoms questionnaires, nasal inhalation flow readings during the in-person visits at the hospital. Investigators will also attempt to mimic allergen and pollution exposures, and track how the treatment affects one's nasal responses during visits. On days where participants do not have in-person visits, participants will continue using the treatment product on a daily basis. After one cycle of treatment, participants will go through a wash-out period before starting the second cycle with the opposite treatment (Budesonide (Rhinocort)/placebo).

Investigators are not expecting that participants' responses to the treatments or exposures will be noticeable to the participants. Any responses that may occur will probably only be detectable through careful examination of the collected nasal samples on a genetic basis. However, being able to understand the subtle changes will help investigators optimize and better understand the use of these treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18 - 65 years. (Female subjects must be postmenopausal, surgically sterile or using medically accepted contraceptive means, as judged by the investigator).
* Asymptomatic subjects (not experiencing rhinitis symptoms at the time of screening).
* A clinical diagnosis of allergic rhinitis (dust mite, grass mix or tree mix) for at least the previous two years.
* Subjects with a need of treatment for their nasal symptoms during the pollen season of such severity that it required pharmacological therapy each year for the last two consecutive years.
* Willingness to participate as indicated by a signed informed consent. Signed consent must be obtained from the subject prior to start of any study-related procedures.
* Availability and ability for all planned site visits
* A nasal allergen challenge resulting in at least five sneezes and/or a recorded score of >2 in either nasal obstruction or runny nose

Exclusion Criteria:

* Subjects with confirmed hypersensitivity to budesonide.
* Subjects with previous or current respiratory- cardiovascular-, renal-, liver-, endocrinological or other diseases or conditions which may influence the subject's participation in the study or the result hereof, as judged by the investigator.
* Subjects with a planned hospitalization or planned blood-donation during the study.
* Women who are pregnant or nursing.
* Diseases or conditions which might interfere with the evaluation of efficacy and safety:
* Subjects with structural abnormalities of the nose (e.g. septal deviation, nasal polyps) or other diseases (infectious rhinitis, sinusitis, rhinitis medicamentosa and atrophic or non- allergic rhinitis) which could cause significant nasal obstruction or other symptoms which could have any significant influence on the investigated disease as judged by the investigator.
* History of asthma.
* PAR (with an exception, see inclusion criterion 3).
* Subjects allergic to other allergens occurring during the study period.
* Systemic corticosteroid use within 2 months, topical corticosteroid use within 2 weeks, antihistamine use within 1 week, leukotriene antagonist use within one week or immunotherapy within 2 years of baseline visit (or stop at screening)
* Upper respiratory infection within 2 weeks of baseline visit
* Use of tobacco within 1 year of baseline
* Chronic medical condition that could interfere with evaluation of rhinitis endpoints (e.g. allergic skin conditions, active infections, asthma, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Budesonide affect on allergic rhinitis plus allergen (48 hrs) | Baseline vs 48 hours
  Change in DNA methylation in the budesonide group compared with placebo.
  DNA methylation measurement tool:
  Illumina Infinium MethylationEPIC BeadChip (interrogates 866,895 CpG sites across the human genome)
  Unit of Measure:
  For each targeted CpG site, the intensity of fluorescence will be translated into a level of DNA methylation which is either represented as a β value, a number between 0 and 1 (0 = no methylated, 1 = fully methylated) for visualization and interpretation, or a logit-transformed β value "M value" for statistical analysis.

SECONDARY OUTCOMES:
Budesonide affect on allergic rhinitis plus allergen (24 hrs) | Baseline vs 24 hours
  Change in DNA methylation in the budesonide group compared with placebo.
  DNA methylation measurement tool:
  Illumina Infinium MethylationEPIC BeadChip (interrogates 866,895 CpG sites across the human genome)
  Unit of Measure:
  For each targeted CpG site, the intensity of fluorescence will be translated into a level of DNA methylation which is either represented as a β value, a number between 0 and 1 (0 = no methylated, 1 = fully methylated) for visualization and interpretation, or a logit-transformed β value "M value" for statistical analysis.
Budesonide affect on allergic rhinitis plus pollution (48 hrs) | Baseline vs 48 hours
  Change in DNA methylation in the budesonide group compared with placebo.
  DNA methylation measurement tool:
  Illumina Infinium MethylationEPIC BeadChip (interrogates 866,895 CpG sites across the human genome)
  Unit of Measure:
  For each targeted CpG site, the intensity of fluorescence will be translated into a level of DNA methylation which is either represented as a β value, a number between 0 and 1 (0 = no methylated, 1 = fully methylated) for visualization and interpretation, or a logit-transformed β value "M value" for statistical analysis.
Budesonide affect on allergic rhinitis plus pollution (24 hrs) | Baseline vs 24 hours
  Change in DNA methylation in the budesonide group compared with placebo.
  DNA methylation measurement tool:
  Illumina Infinium MethylationEPIC BeadChip (interrogates 866,895 CpG sites across the human genome)
  Unit of Measure:
  For each targeted CpG site, the intensity of fluorescence will be translated into a level of DNA methylation which is either represented as a β value, a number between 0 and 1 (0 = no methylated, 1 = fully methylated) for visualization and interpretation, or a logit-transformed β value "M value" for statistical analysis.
Change in Total Nasal Symptoms Score (TNSS) (30 min) | Baseline vs 30-minute post allergen challenge
  Change from allergen baseline in Total Nasal Symptoms Score (TNSS) in the budesonide group compared with placebo 30 minutes after first allergen challenge. TNSS is evaluated on a scale of 0 to 12; with 0 being none and 12 being severe.
Change in Peak Nasal Inspiratory Flow (PNIF) (30 min) | Baseline vs 30-minute post allergen challenge
  Change from allergen baseline in PNIF in the budesonide group compared with placebo 30 minutes after first allergen challenge.
Changes in Concentration of Cytokines | Through study completion, approximately 4 months.
  Change in concentration of cytokines and related protein markers (such as human IL-1 beta, IL-4, IL-6, IL-10, IL-13, TNF-alpha, etc.) across groups and times in the study.
  Cytokine measurement tool:
  Meso Scale Discovery Multiplex and similar ELISA assays that test for the mentioned markers.
  Unit of Measure:
  Concentration (picograms of analyte per ml of undiluted sample) will be calculated from standard curves provided with the assays. Concentration detection ranges between 1-10,000pg/ml. Concentration values will be used for visualization and statistical analysis.

OTHER OUTCOMES:
Change in Total Nasal Symptoms Score (TNSS) (48 hrs) | Baseline vs 48 hours
  Change from allergen baseline Total Nasal Symptoms Score (TNSS) in the budesonide group compared with placebo. TNSS is evaluated on a scale of 0 to 12; with 0 being none and 12 being severe.
Change in Total Nasal Symptoms Score (TNSS) (24 hrs) | Baseline vs 24 hours
  Change from allergen baseline Total Nasal Symptoms Score (TNSS) in the budesonide group compared with placebo. TNSS is evaluated on a scale of 0 to 12; with 0 being none and 12 being severe.
Change in Peak Nasal Inspiratory Flow (PNIF) (48 hrs) | Baseline vs 48 hours
  Change from allergen baseline PNIF in the budesonide group compared with placebo.
Change in Peak Nasal Inspiratory Flow (PNIF) (24 hrs) | Baseline vs 24 hours
  Change from allergen baseline PNIF in the budesonide group compared with placebo.
Comparison of Budesonide vs placebo in the absence of allergen or pollution challenge. | Through study completion, approximately 4 months.
  Change from treatment naïve baseline in DNA methylation attributable to intranasal budesonide compared with placebo in the absence of a nasal allergen or pollution challenge following 14 days of treatment.
  DNA methylation measurement tool:
  Illumina Infinium MethylationEPIC BeadChip (interrogates 866,895 CpG sites across the human genome)
  Unit of Measure:
  For each targeted CpG site, the intensity of fluorescence will be translated into a level of DNA methylation which is either represented as a β value, a number between 0 and 1 (0 = no methylated, 1 = fully methylated) for visualization and interpretation, or a logit-transformed β value "M value" for statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Carlsten, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No